CLINICAL TRIAL: NCT03711227
Title: Procalcitonin at Zero and 24 Hours as a Prognostic Factor in Patients With Pneumonia
Status: Completed | Type: Observational
Sponsor: Corewell Health South (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Sponsor
Other Study IDs: MMMC#1577
Record Dates: First submitted 2018-06-02; First posted 2018-10-18 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2019-10

CONDITIONS: Pneumonia
Keywords: Serial Procalcitonin, Admitted Pneumonia, qSOFA, Sepsis
MeSH Terms: conditions — Pneumonia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Procalcitonin lab test: A procalcitonin order bundle will be created for admitted patients with pneumonia. This prepopulated bundle includes an initial and 24 hour procalcitonin level. These patients will receive treatment for their pneumonia as is deemed appropriate by their care teams, both in the Emergency Department and while an inpatient. Then, after discharge, the 30 day mortality, length of stay, choice of antibiotic therapy, and qSOFA score (which will be retroactively calculated) will be compared to the patient's initial and 24 hour procalcitonin level.
  Interventions: Diagnostic Test: Procalcitonin lab test

INTERVENTIONS:
Diagnostic Test: Procalcitonin lab test — A procalcitonin order bundle will be created for admitted patients with pneumonia. This prepopulated bundle includes an initial and 24 hour procalcitonin level.

SUMMARY:
Procalcitonin levels checked initially and at 24 hours will correlate with disease severity, morbidity, and mortality. Patients who have a higher procalcitonin level initially and at 24 hours will likely have higher qSOFA scores, longer lengths of stay, longer duration of antibiotics and higher 30 day mortality rates.

DETAILED DESCRIPTION:
A procalcitonin order bundle will be created for admitted patients with pneumonia. This prepopulated bundle includes an initial and 24 hour procalcitonin level, much like the current initial and 4 hour lactate orders are set-up. These patients will receive treatment for their pneumonia as is deemed appropriate by their care teams, both in the Emergency Department and while an inpatient. Then, after discharge, the 30 day mortality, length of stay, choice of antibiotic therapy, and qSOFA score (which will be retroactively calculated) will be compared to the patient's initial and 24 hour procalcitonin level.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen at Lakeland St. Joseph and Niles Hospitals in the emergency department and who are then subsequently admitted with pneumonia at Lakeland St. Joseph and Niles Hospitals

Exclusion Criteria:

* Any patients not admitted with pneumonia, any patients who are admitted with another primary diagnosis other than pneumonia, any patients who do not have an initial or 24 hour procalcitonin level result, and any patients less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen at Lakeland St. Joseph and Niles Hospitals in the emergency department and who are then subsequently admitted with pneumonia at Lakeland St. Joseph and Niles Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Procalcitonin level | Measured at baseline and at 24 hours
  Change in procalcitonin level in the blood serum

SECONDARY OUTCOMES:
qSOFA score | baseline and at 24 hours
  qSOFA score is based on blow blood pressure, high respiratory rate, and altered mental status
Length of stay | an average of 30 days
  Length of stay in days, total stay from admission until discharge
Duration of antibiotics | an average of 30 days
  Antibiotic treatment length in days
30 Day Mortality | 30 days
  Number of patients who expire vs those alive at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michelino Mancini, DO, Principal Investigator — Lakeland Hospitals at St. Joseph and Niles
Locations (1):
- Lakeland Regional Healthcare, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD data

REFERENCES:
- [Background] Bloos F, Marshall JC, Dellinger RP, Vincent JL, Gutierrez G, Rivers E, Balk RA, Laterre PF, Angus DC, Reinhart K, Brunkhorst FM. Multinational, observational study of procalcitonin in ICU patients with pneumonia requiring mechanical ventilation: a multicenter observational study. Crit Care. 2011;15(2):R88. doi: 10.1186/cc10087. Epub 2011 Mar 7. PMID 21385367
- [Background] Boussekey N, Leroy O, Alfandari S, Devos P, Georges H, Guery B. Procalcitonin kinetics in the prognosis of severe community-acquired pneumonia. Intensive Care Med. 2006 Mar;32(3):469-72. doi: 10.1007/s00134-005-0047-8. Epub 2006 Feb 14. PMID 16477418
- [Background] Chan YL, Tseng CP, Tsay PK, Chang SS, Chiu TF, Chen JC. Procalcitonin as a marker of bacterial infection in the emergency department: an observational study. Crit Care. 2004 Feb;8(1):R12-20. doi: 10.1186/cc2396. Epub 2003 Nov 20. PMID 14975050
- [Background] Christ-Crain M, Muller B. Procalcitonin and pneumonia: is it a useful marker? Curr Infect Dis Rep. 2007 May;9(3):233-40. doi: 10.1007/s11908-007-0037-9. PMID 17430706
- [Background] Garnacho-Montero J, Huici-Moreno MJ, Gutierrez-Pizarraya A, Lopez I, Marquez-Vacaro JA, Macher H, Guerrero JM, Puppo-Moreno A. Prognostic and diagnostic value of eosinopenia, C-reactive protein, procalcitonin, and circulating cell-free DNA in critically ill patients admitted with suspicion of sepsis. Crit Care. 2014 Jun 5;18(3):R116. doi: 10.1186/cc13908. PMID 24903083
- [Background] Hicks CW, Engineer RS, Benoit JL, Dasarathy S, Christenson RH, Peacock WF. Procalcitonin as a biomarker for early sepsis in the emergency department. Eur J Emerg Med. 2014 Apr;21(2):112-7. doi: 10.1097/MEJ.0b013e328361fee2. PMID 23669296
- [Background] Huang DT, Weissfeld LA, Kellum JA, Yealy DM, Kong L, Martino M, Angus DC; GenIMS Investigators. Risk prediction with procalcitonin and clinical rules in community-acquired pneumonia. Ann Emerg Med. 2008 Jul;52(1):48-58.e2. doi: 10.1016/j.annemergmed.2008.01.003. Epub 2008 Mar 17. PMID 18342993
- [Background] Kim SY, Jeong TD, Lee W, Chun S, Min WK. Procalcitonin in the assessment of bacteraemia in emergency department patients: results of a large retrospective study. Ann Clin Biochem. 2015 Nov;52(Pt 6):654-9. doi: 10.1177/0004563214568685. Epub 2015 Jan 9. PMID 25575698
- [Background] Le Bel J, Hausfater P, Chenevier-Gobeaux C, Blanc FX, Benjoar M, Ficko C, Ray P, Choquet C, Duval X, Claessens YE; ESCAPED study group. Diagnostic accuracy of C-reactive protein and procalcitonin in suspected community-acquired pneumonia adults visiting emergency department and having a systematic thoracic CT scan. Crit Care. 2015 Oct 16;19:366. doi: 10.1186/s13054-015-1083-6. PMID 26472401
- [Background] Lipinska-Gediga M, Mierzchala-Pasierb M, Durek G. Procalcitonin kinetics - prognostic and diagnostic significance in septic patients. Arch Med Sci. 2016 Feb 1;12(1):112-9. doi: 10.5114/aoms.2016.57587. Epub 2016 Feb 2. PMID 26925126
- [Background] Liu D, Su LX, Guan W, Xiao K, Xie LX. Prognostic value of procalcitonin in pneumonia: A systematic review and meta-analysis. Respirology. 2016 Feb;21(2):280-8. doi: 10.1111/resp.12704. Epub 2015 Dec 10. PMID 26662169
- [Background] Masia M, Gutierrez F, Shum C, Padilla S, Navarro JC, Flores E, Hernandez I. Usefulness of procalcitonin levels in community-acquired pneumonia according to the patients outcome research team pneumonia severity index. Chest. 2005 Oct;128(4):2223-9. doi: 10.1378/chest.128.4.2223. PMID 16236878
- [Background] Meisner M, Tschaikowsky K, Palmaers T, Schmidt J. Comparison of procalcitonin (PCT) and C-reactive protein (CRP) plasma concentrations at different SOFA scores during the course of sepsis and MODS. Crit Care. 1999;3(1):45-50. doi: 10.1186/cc306. PMID 11056723
- [Background] Park JH, Wee JH, Choi SP, Oh SH. The value of procalcitonin level in community-acquired pneumonia in the ED. Am J Emerg Med. 2012 Sep;30(7):1248-54. doi: 10.1016/j.ajem.2011.08.009. Epub 2011 Oct 24. PMID 22030193
- [Background] Pfister R, Kochanek M, Leygeber T, Brun-Buisson C, Cuquemelle E, Machado MB, Piacentini E, Hammond NE, Ingram PR, Michels G. Procalcitonin for diagnosis of bacterial pneumonia in critically ill patients during 2009 H1N1 influenza pandemic: a prospective cohort study, systematic review and individual patient data meta-analysis. Crit Care. 2014 Mar 10;18(2):R44. doi: 10.1186/cc13760. PMID 24612487
- [Background] Schuetz P, Amin DN, Greenwald JL. Role of procalcitonin in managing adult patients with respiratory tract infections. Chest. 2012 Apr;141(4):1063-1073. doi: 10.1378/chest.11-2430. PMID 22474148
- [Background] Schuetz P, Birkhahn R, Sherwin R, Jones AE, Singer A, Kline JA, Runyon MS, Self WH, Courtney DM, Nowak RM, Gaieski DF, Ebmeyer S, Johannes S, Wiemer JC, Schwabe A, Shapiro NI. Serial Procalcitonin Predicts Mortality in Severe Sepsis Patients: Results From the Multicenter Procalcitonin MOnitoring SEpsis (MOSES) Study. Crit Care Med. 2017 May;45(5):781-789. doi: 10.1097/CCM.0000000000002321. PMID 28257335
- [Background] Schuetz P, Maurer P, Punjabi V, Desai A, Amin DN, Gluck E. Procalcitonin decrease over 72 hours in US critical care units predicts fatal outcome in sepsis patients. Crit Care. 2013 Jun 20;17(3):R115. doi: 10.1186/cc12787. PMID 23787145
- [Background] Shi Y, Peng JM, Hu XY, Wang Y. The utility of initial procalcitonin and procalcitonin clearance for prediction of bacterial infection and outcome in critically ill patients with autoimmune diseases: a prospective observational study. BMC Anesthesiol. 2015 Oct 7;15:137. doi: 10.1186/s12871-015-0122-9. PMID 26446077
- [Background] Shomali W, Hachem R, Chaftari AM, Jiang Y, Bahu R, Jabbour J, Raad S, Al Shuaibi M, Al Wohoush I, Raad I. Can procalcitonin distinguish infectious fever from tumor-related fever in non-neutropenic cancer patients? Cancer. 2012 Dec 1;118(23):5823-9. doi: 10.1002/cncr.27602. Epub 2012 May 17. PMID 22605389
- [Background] Trasy D, Tanczos K, Nemeth M, Hankovszky P, Lovas A, Mikor A, Laszlo I, Hajdu E, Osztroluczki A, Fazakas J, Molnar Z; EProK study group. Early procalcitonin kinetics and appropriateness of empirical antimicrobial therapy in critically ill patients: A prospective observational study. J Crit Care. 2016 Aug;34:50-5. doi: 10.1016/j.jcrc.2016.04.007. Epub 2016 Apr 13. PMID 27288610
- [Background] Wang XJ, Tan TT, Lim ST, Farid M, Tao M, Quek R, Chan A, Tang T. Role of Procalcitonin in Differentiating between Infectious and Noninfectious Fevers among Patients with Lymphoma. Pharmacotherapy. 2017 Aug;37(8):908-915. doi: 10.1002/phar.1963. Epub 2017 Jul 18. PMID 28556122